CLINICAL TRIAL: NCT03924557
Title: A Randomized Pragmatic Trial of Genotype-guided Supportive Care in Symptom Treatment of Cancer Patients
Brief Title: Genotype-guided Supportive Care in Symptom Treatment of Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding issues
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UF-ETG-002; OCR20388 (Other: UF OnCore); IRB201901177 (Other: University of Florida)
Record Dates: First submitted 2019-04-19; First posted 2019-04-23 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Chemotherapy; Supportive Care; Genotyping

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, parallel arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genotyping Intervention Supportive Care (Active Comparator): For those randomized to the genotype intervention group, genotype results will be returned in the EHR pre-emptively and supportive care will be prescribed based on genotype results.
  Interventions: Diagnostic Test: Genotype-guided Supportive Care
- Delayed Genotyping Intervention Supportive Care (No Intervention): For those randomized to the delayed genotype intervention group, supportive care will be prescribed based on usual clinical practice.

INTERVENTIONS:
Diagnostic Test: Genotype-guided Supportive Care — In this arm, supportive care will be administered based on the results of the genotype test.
  Arms: Genotyping Intervention Supportive Care

SUMMARY:
Cancer patients often require administration of multiple supportive care pharmacotherapies while receiving chemotherapy regardless the type of cancer. Supportive care therapies are commonly prescribed to nearly all cancer patients and could include antiemetics (ondansetron), pain management (opiates), GI protection (PPIs), antidepressants (select SSRIs), anticoagulation (warfarin) and antifungal prophylaxis (voriconazole). These are all are associated with known pharmacogenetic interactions, which in some cases render the drugs ineffective or toxic. This could result in negative impacts on quality of life in patients who are already undergoing complicated and costly anticancer regimens. Pharmacogenetic-guided therapy based on an individual patient's genetic profile could potentially target symptoms for which an individual is uniquely susceptible, guiding use of medications that are most likely to be effective, thereby reducing unnecessary physical complications and financial strain. It is hypothesized that patients in the genotype intervention arm will report lower scores for overall symptom distress as compared to patients in the delayed genotype intervention arm following initiation of chemotherapy.

DETAILED DESCRIPTION:
This is a single center, pilot randomized pragmatic clinical trial (PCT) of 500 cancer patients who are undergoing chemotherapy for newly diagnosed or recurrent cancers. Patients will be randomized to genotyping intervention vs delayed genotyping intervention supportive care. Supportive care regimens may include therapies for antiemesis (ondansetron), pain management (opiates), GI protection (PPIs), antidepressants (select SSRIs), and antifungal prophylaxis (voriconazole), and warfarin depending on their chemotherapy regimen.

For those randomized to the genotype intervention group, genotype results will be returned in the EHR pre-emptively and supportive care will be prescribed based on genotype results. For those randomized to the delayed genotype intervention group, supportive care will be prescribed based on usual clinical practice. Both groups will be followed for 3 months and undergo assessments with the MDASI questionnaire four times (pre-chemotherapy, and 2 weeks, 4 weeks and 12 weeks post initiation of chemotherapy.

Records for patients receiving outpatient care at the UF Health Cancer Center clinic at the Medical Plaza will be screened based on inclusion / exclusion criteria for participation in this study. Those that meet criteria will be offered participation. Participation is expected to last approximately 12 weeks and the study will be open for 30-36 months.

ELIGIBILITY:
Inclusion Criteria:

* Must have a clinical diagnosis of solid tumor cancer and be seeking treatment and supportive care at the UF Health Cancer Center (Medical Plaza)
* Patients must plan to receive chemotherapy known to be associated with the need for supportive care within 30 days of enrollment
* Life expectancy must be greater than 6 months
* Must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Written informed consent obtained from the patient
* The ability for the patient to comply with all the study-related procedures.

Exclusion Criteria:

* Patients unwilling or unable to provide voluntary informed consent
* Patients who are unwilling or unable to comply with protocol requirement and/or follow-up procedures
* Patients planned to undergo cancer therapy other than chemotherapy (i.e., radiation, surgery or hormonal treatment alone)
* Prisoners or patients who are involuntarily incarcerated. Patients who are compulsorily detained for treatment of either a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Change in patient MDASI scoring | At pre-chemotherapy (baseline), 2 weeks, 4 weeks, and 12 weeks post initiation of chemotherapy.
  The M. D. Anderson Symptom Inventory (MDASI) is a multisymptom patient-reported outcome measure. Participants are asked to recall symptom interference and severity during the past 24 hours and rate the symptom using a numeric rating scale, 0-10. For the symptom interference questions, 10 means interfered completely and 0 is did not interfere. For the symptom severity questions, 10 means as bad as you can imagine and 0 is not present. The MDASI questionnaire will evaluate symptom distress and core symptoms of patients at four separate time points.

SECONDARY OUTCOMES:
Change in patient medication use | At pre-chemotherapy (baseline), 2 weeks, 4 weeks, and 12 weeks post initiation of chemotherapy.
  Concomitant Medication Review will be collected from patients or from their electronic medical record to evaluate differences in medication use (drug and dose) based on randomized group.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Cooper-DeHoff, Pharm D, MS, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health at the University of Florida, Gainesville, Florida
  - UF Health Cancer Center, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cicali EJ, Eddy E, Gong Y, Elchynski AL, Pena Del Aguila K, Basha T, Daily KC, Dickson L, Fischer S, Hastings-Monari E, Jones D Jr, Ramnaraign BH, DeRemer DL, George TJ, Cooper-DeHoff RM. Implementation of a pharmacogenetic panel-based test for pharmacotherapy-based supportive care in an adult oncology clinic. Clin Transl Sci. 2024 Jul;17(7):e13890. doi: 10.1111/cts.13890. PMID 39046302